CLINICAL TRIAL: NCT02892409
Title: A Phase 1, Double-Blind, Parallel Group Study to Evaluate the Safety and Pharmacokinetics of Quadruple Therapy (Bismuth, Clarithromycin, and Amoxicillin) With TAK-438 Versus Quadruple Therapy With Lansoprazole
Brief Title: TAK-438 Bismuth Drug Interaction Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TAK-438_115; U1111-1179-5816 (Other: WHO); 02892409 (Registry Identifier: ClinicalTrials.gov)
Record Dates: First submitted 2016-09-02; First posted 2016-09-08 (Estimated); Results first posted 2019-01-03 (Actual); Last update posted 2019-01-03 (Actual); Status verified 2018-06

CONDITIONS: Helicobacter Pylori
Keywords: Drug Therapy
MeSH Terms: interventions — Clarithromycin; Amoxicillin; bismuth tripotassium dicitrate; Lansoprazole; 1-(5-(2-fluorophenyl)-1-(pyridin-3-ylsulfonyl)-1H-pyrrol-3-yl)-N-methylmethanamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Clarithromycin + Amoxicillin + Bismuth + Lansoprazole (Active Comparator): Clarithromycin 500 milligram (mg), tablets, orally, twice daily, along with amoxicillin 1000 mg capsules, orally, twice daily, tripotassium bismuth dicitrate 600 mg, tablets, orally, twice daily, and lansoprazole 30 mg, capsules, orally, twice daily on Days 1 to 14.
  Interventions: Drug: Clarithromycin; Drug: Amoxicillin; Drug: Tripotassium bismuth dicitrate; Drug: Lansoprazole
- Clarithromycin + Amoxicillin + Bismuth + TAK-438 (Experimental): Clarithromycin 500 mg, tablets, orally, twice daily, along with amoxicillin 1000 mg, capsules, orally, twice daily, tripotassium bismuth dicitrate 600 mg, tablets, orally, twice daily, and TAK-438 20 mg, tablets, orally, twice daily on Days 1 to 14.
  Interventions: Drug: Clarithromycin; Drug: Amoxicillin; Drug: Tripotassium bismuth dicitrate; Drug: TAK-438

INTERVENTIONS:
Drug: Clarithromycin — Clarithromycin tablets
Drug: Amoxicillin — Amoxicillin capsules
Drug: Tripotassium bismuth dicitrate — Tripotassium bismuth dicitrate tablets
Drug: Lansoprazole — Lansoprazole capsules
  Arms: Clarithromycin + Amoxicillin + Bismuth + Lansoprazole
Drug: TAK-438 — TAK-438 tablets
  Arms: Clarithromycin + Amoxicillin + Bismuth + TAK-438

SUMMARY:
To evaluate the safety, tolerability, and pharmacokinetics (PK) of quadruple therapy with bismuth, clarithromycin, amoxicillin, and TAK-438 versus quadruple therapy with bismuth, clarithromycin, amoxicillin, and lansoprazole.

DETAILED DESCRIPTION:
This is a phase 1, double-blind, parallel group study in participants with Helicobacter pylori (HP positive) who are, additionally, cytochrome P-450 (CYP)2C19 extensive metabolizers (EM) to evaluate the safety, tolerability and pharmacokinetics (PK) of a quadruple therapy with bismuth, clarithromycin, amoxicillin, and TAK-438 versus quadruple therapy with bismuth, clarithromycin, amoxicillin, and lansoprazole. The study will enroll 30 participants.

The treatment phase consists of quadruple therapy twice daily (BID) with tripotassium bismuth dicitrate (600 mg), clarithromycin (500 mg), amoxicillin (1000 mg), and TAK-438 (20 mg) (Group B) or quadruple therapy BID with tripotassium bismuth dicitrate (600 mg), clarithromycin (500 mg), amoxicillin (1000 mg),and lansoprazole (30 mg) (Group A) from Days 1 to 14. Participants will be discharged on Day 15 after final PK blood samples are collected and all procedures performed.

This single-center will be conducted in Korea. Participants will remain confined to the study site from check-in (Day -1) through Day 15 and will followed up through call on Day 17 and return on Day 42 for a follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

1. HP positive participants.
2. Has body mass index between greater than (>) 18 and less than equal to (<=) 30 kilogram per square meter (kg/m^2) and weighs greater than equal to (>=) 50 kilogram (kg).
3. Is willing to abstain from strenuous exercise from 72 hours before first dose (Day 1) until the Follow-up call on Day 17.

Exclusion Criteria:

1. Has a positive urine drug result for drugs of abuse at Screening or Check-in (Day -1).
2. Has a history of drug abuse (defined as any illicit drug use) or a history of alcohol abuse (defined as regular consumption of 21 units or more units per week) at any time prior to the Screening Visit or is unwilling to agree to abstain from alcohol and drugs throughout the study (up to Day 17).
3. Has history of gastroesophageal reflux disease (GERD), symptomatic GERD, erosive esophagitis, duodenal ulcer, gastric ulcer, Barrett's esophagus, or Zollinger-Ellison syndrome.
4. Has undergone therapeutic upper gastrointestinal endoscopic therapy (example, endoscopic hemostasis or excision including biopsy) within 30 days prior to Screening.
5. Has undergone major surgical procedures within the past 1 month or are scheduled to undergo surgical procedures that may affect gastric acid secretion (example, abdominal surgery, vagotomy, or craniotomy).
6. Has a history of cancer, except basal cell carcinoma or Stage 1 squamous cell carcinoma of the skin that has been in remission for at least 5 years prior to Day 1.
7. Has a positive test result for hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibody, human immunodeficiency virus (HIV) antibody/antigen at Screening.
8. Has used nicotine-containing products (including but not limited to cigarettes, pipes, cigars, chewing tobacco, nicotine patch or nicotine gum) within 6 weeks prior to Check-in. Cotinine test is positive at Screening or Check-in.
9. Has poor peripheral venous access. Has donated or lost 450 milliliter (mL) or more of his blood volume (including plasmapheresis), or had a transfusion of any blood product within 90 days prior to Day 1.
10. Has abnormal Screening or Check-in laboratory values that suggest a clinically significant underlying disease or subject with the following laboratory abnormalities: alanine aminotransferase (ALT), aspartate aminotransferase (AST) or total bilirubin > the upper limit of normal (ULN).
11. Has reduced renal function assessed by having an estimated glomerular filtration rate <90 milliliter per min per 1.73 square meter (mL/min/1.73 m^2) (as estimated by Chronic Kidney Disease-Epidemology Collaboration) at Screening or Check-in.

Ages: 19 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2016-09-05 (Actual); Primary Completion 2017-04-17 (Actual); Study Completion 2017-05-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda
Locations (1):
- Seoul, South Korea

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 1 investigative site in Korea from 05 September 2016 to 11 May 2017.
Pre-assignment Details: Participants with diagnosis of positive helicobacter pylori (HP) were enrolled in 1 of the 2 treatment groups to receive: Clarithromycin + Amoxicillin + Tripotassium Bismuth Dicitrate (Bismuth) + Lansoprazole twice daily or Clarithromycin + Amoxicillin + Bismuth + TAK-438 twice daily.
Groups:
- Clarithromycin + Amoxicillin + Bismuth + TAK-438: Clarithromycin 500 milligram (mg), tablets, orally, twice daily, amoxicillin 1000 mg, capsules, orally, twice daily, bismuth 600 mg, tablets, orally, twice daily, and TAK-438 20 mg, tablets, orally, twice daily on Days 1 to 14.
- Clarithromycin + Amoxicillin + Bismuth + Lansoprazole: Clarithromycin 500 mg, tablets, orally, twice daily, amoxicillin 1000 mg capsules, orally, twice daily, bismuth 600 mg, tablets, orally, twice daily, and lansoprazole 30 mg, capsules, orally, twice daily on Days 1 to 14.
Period: Overall Study
Arm/Group | Clarithromycin + Amoxicillin + Bismuth + TAK-438 | Clarithromycin + Amoxicillin + Bismuth + Lansoprazole
Started | 15 | 15
Completed | 12 | 14
Not Completed | 3 | 1
Not completed — Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 2 | 1

BASELINE CHARACTERISTICS:
Population: The safety analysis set included all participants who received at least one dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Clarithromycin + Amoxicillin + Bismuth + TAK-438 | Clarithromycin + Amoxicillin + Bismuth + Lansoprazole | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.8 (6.87) | 33.3 (8.61) | 33.1 (7.66)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 14 | 14 | 28
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 15 | 15 | 30
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Height [Mean (Standard Deviation); unit: centimeter (cm)] | 173.7 (5.04) | 168.9 (5.14) | 171.3 (5.56)
Weight [Mean (Standard Deviation); unit: kilogram (kg)] | 72.41 (5.028) | 66.05 (8.395) | 69.23 (7.528)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilogram per square meter (kg/m^2)] | 24.03 (1.795) | 23.13 (2.271) | 23.58 (2.064)
Smoking Classification [Count of Participants; unit: Participants]
  Never smoked | 14 | 12 | 26
  Ex-smoker | 1 | 3 | 4
Alcohol Consumption [Count of Participants; unit: Participants]
  Drank a couple of days per week | 2 | 0 | 2
  Drank a couple of days per month | 4 | 6 | 10
  Never Drank | 9 | 9 | 18
Caffeine Consumption [Count of Participants; unit: Participants]
  Had caffeine consumption | 7 | 13 | 20
  Had no caffeine consumption | 8 | 2 | 10
Cytochrome P450 2C19 (CYP2C19) Genotype [Count of Participants; unit: Participants]
  *1/*1 | 5 | 6 | 11
  *1/*2 | 6 | 5 | 11
  *1/*3 | 3 | 3 | 6
  *2/*2 | 0 | 0 | 0
  *2/*3 | 1 | 0 | 1
  *3/*3 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Experience at Least One Treatment Emergent Adverse Event (TEAE)
Time Frame: Baseline up to Day 17
Population: The safety analysis set included all participants who received at least one dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Clarithromycin + Amoxicillin + Bismuth + TAK-438 | Clarithromycin + Amoxicillin + Bismuth + Lansoprazole
Number analyzed (Participants) | 15 | 15
percentage of participants | 53.3 | 66.7

2. Primary Outcome: Percentage of Participants Who Discontinue Due to an Adverse Event (AE)
Time Frame: Baseline up to Day 17
Population: The safety analysis set included all participants who received at least one dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Clarithromycin + Amoxicillin + Bismuth + TAK-438 | Clarithromycin + Amoxicillin + Bismuth + Lansoprazole
Number analyzed (Participants) | 15 | 15
percentage of participants | 6.7 | 0.0

3. Primary Outcome: Percentage of Participants Who Meet the Markedly Abnormal Criteria for Safety Laboratory Tests at Least Once Post-dose
Time Frame: Baseline up Day 15
Population: The safety analysis set included all participants who received at least one dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Clarithromycin + Amoxicillin + Bismuth + TAK-438 | Clarithromycin + Amoxicillin + Bismuth + Lansoprazole
Number analyzed (Participants) | 15 | 15
percentage of participants
  Amylase (greater than [>] 2*upper limit of normal) | 0.0 | 6.7
  Potassium (>6.0 millimole per liter [mmol/L]) | 0.0 | 6.7

4. Primary Outcome: Percentage of Participants Who Meet the Markedly Abnormal Criteria for Vital Sign Measurements at Least Once Post-dose
Time Frame: Baseline up to Day 15
Population: The safety analysis set included all participants who received at least one dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Clarithromycin + Amoxicillin + Bismuth + TAK-438 | Clarithromycin + Amoxicillin + Bismuth + Lansoprazole
Number analyzed (Participants) | 15 | 15
percentage of participants
  Body temperature (less than [<] 35.6 celsius [C]) | 0.0 | 6.7
  Body temperature (>37.7 C) | 6.7 | 6.7
  Systolic blood pressure(<85 millimeter of mercury) | 6.7 | 6.7
  Diastolic blood pressure(<50millimeter of mercury) | 6.7 | 6.7

5. Primary Outcome: Percentage of Participants Who Meet the Markedly Abnormal Criteria for Safety Electrocardiogram (ECG) Parameters at Least Once Post-dose
Time Frame: Baseline up to Day 15
Population: The safety analysis set included all participants who received at least one dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Clarithromycin + Amoxicillin + Bismuth + TAK-438 | Clarithromycin + Amoxicillin + Bismuth + Lansoprazole
Number analyzed (Participants) | 15 | 15
percentage of participants | 0.0 | 6.7

6. Primary Outcome: Cmax: Maximum Observed Plasma Concentration for Bismuth
Time Frame: Day 14 pre-dose and at multiple timepoints (up to 12 hours) post-dose
Population: The pharmacokinetic (PK) analysis set included all participants who received study drug, had sufficient plasma/urine concentration data to calculate at least one PK parameter, and had no significant protocol deviations.
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Clarithromycin + Amoxicillin + Bismuth + TAK-438 | Clarithromycin + Amoxicillin + Bismuth + Lansoprazole
Number analyzed (Participants) | 12 | 14
nanogram per milliliter (ng/mL) | 28.08 (11.691) | 30.14 (24.612)
Statistical Analysis 1: Comparison: Clarithromycin + Amoxicillin + Bismuth + TAK-438 vs Clarithromycin + Amoxicillin + Bismuth + Lansoprazole; Test type: Equivalence — LS Mean Ratio (TAK-438/Lansoprazole), 95 percent (%) confidence interval (CI) of the ratio were obtained by taking the anti-log of the difference or confidence limits of difference between the LS means of test and reference on the natural logarithmic scale; Least Square (LS) Mean Ratio = 105.1, 95% CI 2-sided [66.051 to 167.183]

7. Primary Outcome: AUCτ: Area Under the Plasma Concentration-time Curve From Time 0 to Time Tau Over the Dosing Interval for Bismuth
Time Frame: Day 14 pre-dose and at multiple timepoints (up to 12 hours) post-dose
Population: The PK analysis set included all participants who received study drug, had sufficient plasma/urine concentration data to calculate at least one PK parameter, and had no significant protocol deviations.
Measure: Mean (Standard Deviation); unit: hours nanogram per milliliter (h*ng/mL)
Arm/Group | Clarithromycin + Amoxicillin + Bismuth + TAK-438 | Clarithromycin + Amoxicillin + Bismuth + Lansoprazole
Number analyzed (Participants) | 12 | 14
hours nanogram per milliliter (h*ng/mL) | 103.0 (37.498) | 111.1 (45.010)
Statistical Analysis 1: Comparison: Clarithromycin + Amoxicillin + Bismuth + TAK-438 vs Clarithromycin + Amoxicillin + Bismuth + Lansoprazole; Test type: Equivalence — LS Mean Ratio (TAK-438/Lansoprazole), 95% CI of the ratio were obtained by taking the anti-log of the difference or confidence limits of difference between the LS means of test and reference on the natural logarithmic scale; LS Mean Ratio = 93.6, 95% CI 2-sided [67.137 to 130.569]

8. Primary Outcome: Aeτ: Amount of Drug Excreted in Urine During a Dosing Interval for Bismuth
Time Frame: Day 14 pre-dose and at multiple timepoints (up to 12 hours) post-dose
Population: The PK analysis set included all participants who received study drug, had sufficient plasma/urine concentration data to calculate at least one PK parameter, and had no significant protocol deviations. The PK analysis set where data was available at specified timepoints.
Measure: Mean (Standard Deviation); unit: nanogram (ng)
Arm/Group | Clarithromycin + Amoxicillin + Bismuth + TAK-438 | Clarithromycin + Amoxicillin + Bismuth + Lansoprazole
Number analyzed (Participants) | 12 | 13
nanogram (ng) | 497300 (202270) | 537600 (188340)

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events are adverse events that started after the first dose of double-blind study drug and up to Day 17
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Clarithromycin + Amoxicillin + Bismuth + TAK-438 | Clarithromycin + Amoxicillin + Bismuth + Lansoprazole
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 8/15 | 10/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Clarithromycin + Amoxicillin + Bismuth + TAK-438 (N=15) | Clarithromycin + Amoxicillin + Bismuth + Lansoprazole (N=15)
Palpitations (Cardiac disorders) | 1 | 0
Hyperthyroidism (Endocrine disorders) | 1 | 0
Eye pruritus (Eye disorders) | 0 | 1
Faeces discoloured (Gastrointestinal disorders) | 1 | 2
Diarrhoea (Gastrointestinal disorders) | 1 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1
Infrequent bowel movements (Gastrointestinal disorders) | 1 | 0
Feeling hot (General disorders) | 2 | 1
Catheter site erythema (General disorders) | 0 | 1
Chest discomfort (General disorders) | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Laceration (Injury, poisoning and procedural complications) | 1 | 0
Neutrophil count decreased (Investigations) | 0 | 1
Dysgeusia (Nervous system disorders) | 0 | 3
Dizziness (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Menstruation irregular (Reproductive system and breast disorders) | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 3 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Research Organization shall not publish any articles or papers nor make any presentations, nor assist any other person in publishing any articles or papers or in making any presentations relating or referring to the Study or any results, data or insights from or any data, information or materials obtained or generated in the performance of its obligations without the prior written consent of Takeda, which consent may be granted or withheld in Takeda's sole discretion.

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-05-15): https://cdn.clinicaltrials.gov/large-docs/09/NCT02892409/SAP_000.pdf
  • Study Protocol (2016-11-21): https://cdn.clinicaltrials.gov/large-docs/09/NCT02892409/Prot_001.pdf